CLINICAL TRIAL: NCT04304807
Title: Effect of Melatonin on Feeding Intolerance and Incidence of Necrotizing Enterocolitis in Preterm Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona Mostafa El-Gammall, Resident of pediatrics and neonatology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PediatricsASU
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Preterm Infant; Feeding Intolerance; Necrotizing Enterocolitis
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Forty five preterm infants with signs of feeding intolerance who received 20 mg of melatonin treatment in addition to traditional antibiotic treatment.
  Interventions: Drug: Melatonin 20 mg
- Group II (Sham Comparator): Forty five preterm infants with signs of feeding intolerance who received traditional antibiotic treatment only.
  Interventions: Drug: Traditional antibiotic treatment

INTERVENTIONS:
Drug: Melatonin 20 mg — Melatonin was given as a total dose of 20 mg via enteral route in two doses of 10 mg each with a 1 hour interval in between.
  Other Names: Melatonin treatment
  Arms: Group I
Drug: Traditional antibiotic treatment — Traditional antibiotic treatment was given to both groups with feeding intolerance according to treatment protocols by neonatal intensive care units of Ain Shams University
  Other Names: Conventional treatment
  Arms: Group II

SUMMARY:
Assesses the efficacy of melatonin in treatment of feeding intolerance in preterm infants, the time needed to reach full enteral intake, the incidence of necrotizing enterocolitis and measures the level of tumor necrosis factor-alpha as a marker of oxidative stress.

DETAILED DESCRIPTION:
This is a prospective study held on ninety preterm infants in Ain Shams University neonatal intensive care units. All enrolled neonates were suffering from feeding intolerance in the form of abdominal distension, gastric residuals or bloody stools. The first group of forty five infants were given melatonin in addition to traditional antibiotic treatment. The second group of forty five infants were given traditional antibiotic treatment only. Both groups were followed up clinically as regards improvement of clinical signs of feeding intolerance and laboratory results till they reached full enteral intake. Both groups were compared as regards incidence of necrotizing enterocolitis and level of tumor necrosis factor-alpha after 72 hours of starting treatment as a marker of oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants (<37 weeks of gestation)
* Evidence of feeding intolerance

Exclusion Criteria:

* Infants with hypoxic ischemic encephalopathy
* Infants on nothing per os
* Infants with high oxygen needs wither on invasive or non-invasive mechanical ventilation
* Major congenital anomalies
* Intracranial hemorrhage
* Respiratory distress syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-12-24 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Melatonin as an antioxidant and free radical scavenger in feeding intolerance in preterm infants | 3 days
  Melatonin efficacy in treatment of oxidative stress in preterm infants with feeding intolerance was assessed by measuring level of tumor necrosis factor- alpha.
Melatonin efficacy in reducing incidence of necrotizing enterocolitis in preterm infants | 1 week
  Melatonin efficacy in reducing incidence of necrotizing enterocolitis by radiological criteria: abdominal ultrasound showing pneumatosis intestinalis.
Effect of melatonin on time needed to reach full enteral intake in preterm infants with feeding intolerance | 2 weeks
  Preterm infants with feeding intolerance were observed for the time needed to reach full enteral intake.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Pediatrics Department, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and informed consent form will be available upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months after finishing the study